CLINICAL TRIAL: NCT00956592
Title: A Randomized Control Trial to Determine First Attempt Intubation Success With the CMAC Laryngoscope vs. Macintosh Blade in Airways Predicted to be Difficult
Brief Title: Clinical Evaluation of the Storz CMAC Laryngoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Michael Aziz, Associate Professor Department of Anesthesiology & Perioperative Medicine, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00003272
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Results first posted 2011-03-09 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Intubation; Airway Management
Keywords: Video laryngoscopy; Intubation success; Difficult airway; CMAC laryngoscope

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CMAC Video laryngoscope (Active Comparator): Subjects will have their intubation attempted first with the CMAC video laryngoscope
  Interventions: Device: CMAC video laryngoscope
- Macintosh blade (Active Comparator): Patients will have their first intubation attempted utilizing the conventional Macintosh design laryngoscope blade
  Interventions: Device: Macintosh laryngoscope

INTERVENTIONS:
Device: CMAC video laryngoscope — Intubation utilizing the assistance of video enhancement
  Other Names: CMAC; Storz laryngoscope
  Arms: CMAC Video laryngoscope
Device: Macintosh laryngoscope — Patients will be intubated utilizing either a Macintosh 3 or Macintosh 4 designed blade
  Other Names: Mac blade
  Arms: Macintosh blade

SUMMARY:
This study aims to evaluate the utility of a video assisted device for intubation (placement of a breathing tube) during surgery. This study specifically aims to compare a video assisted intubation with the CMAC laryngoscope to conventional devices in the setting of intubations predicted to be difficult.

DETAILED DESCRIPTION:
Patients will be specifically screened for predictors by history and physical exam of potential airway difficulty. The role of video laryngoscopy in airways predicted to be difficult is poorly defined. This study aims to recognize if video laryngoscopy is more useful than conventional laryngoscopy as a first attempt for those with anticipated difficulty.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients presenting for elective surgery who are fasted and who have one of the following difficult airway predictors:

  * mallampati classification 3
  * mallampati classification 4
  * Reduced mouth opening (<3cm)
  * reduced cervical motion
  * history of previous difficult intubation or multiple laryngoscopy attempts

Exclusion Criteria:

* Patients less than 18 years old, patients who are not fasted (>6 hrs. NPO)
* Patients who have contraindications to the administration of neuromuscular blocking drugs
* Patients who have a documented history of intubation on first attempt with C-L grade 1 laryngeal view
* Patients who are deemed to difficult and dangerous to anesthetize without first securing an airway.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Aziz, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Jungbauer A, Schumann M, Brunkhorst V, Borgers A, Groeben H. Expected difficult tracheal intubation: a prospective comparison of direct laryngoscopy and video laryngoscopy in 200 patients. Br J Anaesth. 2009 Apr;102(4):546-50. doi: 10.1093/bja/aep013. Epub 2009 Feb 20. PMID 19233881

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at OHSU OR and procedure rooms. 300 patients were enrolled in the study from 10/09-12/10
Pre-assignment Details: 4 exclusions were noted for failure to follow the randomization
Groups:
- CMAC Video Laryngoscope: Subjects will have their intubation attempted first with the CMAC video laryngoscope. Success is measured as confirmed tube placement with single blade insertion
- Macintosh Blade: Patients will have their first intubation attempted utilizing the conventional Macintosh design laryngoscope blade. Success is measured as confirmed tube placement with a single blade insertion
Period: Overall Study
Arm/Group | CMAC Video Laryngoscope | Macintosh Blade
Started | 150 | 150
Completed | 149 | 147
Not Completed | 1 | 3
Not completed — Protocol Violation | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CMAC Video Laryngoscope | Macintosh Blade | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 122 | 114 | 236
  >=65 years | 28 | 36 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (14.2) | 55.4 (14.5) | 54.6 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 65 | 141
  Male | 74 | 85 | 159
Region of Enrollment [Number; unit: participants]
  United States | 150 | 150 | 300

OUTCOME MEASURES:

1. Primary Outcome: Measure of Intubation Success
Description: Success was measured by confirmed tracheal tube placement with one attempt. Any removal of the laryngoscope blade constituted a failure
Time Frame: During each intubation in a 14 month period
Population: 4 patients of the 300 were excluded because the randomization was not followed due to unavailability of equipment or provider preference to remove patient from study
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | CMAC Video Laryngoscope | Macintosh Blade
Number analyzed (Participants) | 149 | 147
Participants | 138 [132 to 144] | 124 [117 to 131]

2. Secondary Outcome: Intubation Time
Description: Time was measured as the duration of laryngoscopy defined by blade insertion to tracheal tube cuff inflation
Time Frame: During laryngoscopy procedure
Population: time
Measure: Mean (90% Confidence Interval); unit: seconds
Arm/Group | CMAC Video Laryngoscope | Macintosh Blade
Number analyzed (Participants) | 149 | 147
seconds | 46 [40 to 51] | 33 [29 to 36]

3. Secondary Outcome: Number of Participants Intubated With a Rescue Device
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | CMAC Video Laryngoscope | Macintosh Blade
Number analyzed (Participants) | 149 | 147
participants | 6 | 12

4. Secondary Outcome: Number of Participants With Complications
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | CMAC Video Laryngoscope | Macintosh Blade
Number analyzed (Participants) | 147 | 149
Participants | 35 | 26

5. Secondary Outcome: Number of Participants With a Laryngeal View Grade of 1 or 2 vs. 3 or 4.
Description: Grade 1= full view of the glottis achieved Grade 2= partial view of the glottis achieved Grade 3= only the epiglottis visualized Grade 4= no laryngeal view achieved
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | CMAC Video Laryngoscope | Macintosh Blade
Number analyzed (Participants) | 149 | 147
Participants
  Grade I view achieved | 103 | 72
  Grade 2 view achieved | 36 | 47
  Grade 3 view achieved | 9 | 26
  Grade 4 view achieved | 1 | 2

6. Secondary Outcome: Number of Particpants Requiring Adjuncts to Assist Intubation
Time Frame: 1 year
Population: Use of bougie or external manipulation
Measure: Count of Participants; unit: Participants
Arm/Group | CMAC Video Laryngoscope | Macintosh Blade
Number analyzed (Participants) | 138 | 124
Participants | 33 | 46

ADVERSE EVENTS:
Arm/Group | CMAC Video Laryngoscope | Macintosh Blade
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/150
Other Adverse Events (participants affected / at risk) | 0/150 | 0/150

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No